CLINICAL TRIAL: NCT04648618
Title: Impact of Obstructive Sleep Apnea on the Expression of Inflammatory Mediators in Diabetic Macular Edema
Brief Title: Obstructive Sleep Apnea and Diabetic Macular Edema Inflammatory Mediators
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Uptown Eye Specialists (Other)
Responsible Party: Sponsor
Other Study IDs: OSA-DME 2
Record Dates: First submitted 2020-11-23; First posted 2020-12-01 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Diabetic Macular Edema; Obstructive Sleep Apnea; Diabetic Retinopathy
Keywords: diabetic macular edema; obstructive sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OSA + DME +: Patients with OSA and DME
- OSA - DME +: Patients with DME, but no evidence of OSA

SUMMARY:
Obstructive sleep apnea (OSA) is characterized by intermittent nocturnal hypoxemia, frequent arousals, fragmented sleep and daytime sleepiness. It has been shown to increase the risk of cardiac and vascular disease through multiple mechanisms including sympathetic hyperactivity, metabolic dysregulation, and activation of oxidative stress and inflammatory pathways.

Diabetic retinopathy is a leading cause of blindness in the working age group, affecting 93 million people worldwide. Diabetic macular edema (DME) is a sight threatening complication and the most common cause of visual loss in patients with diabetes. OSA is frequently associated with diabetes with prevalence ranging from 23 to 86%. However, the relationship between OSA and DME is not well defined. The retina is especially susceptible to hypoxia, being one of the most metabolically active tissues. Many of the same inflammatory mediators have also been found to be elevated in patients with diabetic macular edema, including VEGF, VCAM-1 and IL-6.

There has been no previous study examining the biochemical impact of OSA on patients with DME. We aim to explore this relationship by examining the differences in inflammatory markers expressed in patients with DME who have undergone an overnight sleep study, which is considered the gold standard diagnostic tool in OSA.

DETAILED DESCRIPTION:
The purpose of this study is to compare the levels of inflammatory mediators in diabetic patients with macular edema with and without OSA.

This will be a single centre, prospective, cross-sectional study. We will be recruiting patients undergoing intravitreal injection for diabetic macular edema divided into 2 groups:

* Group 1: diabetic patients with macular edema, no OSA
* Group 2: diabetic patients with macular edema, and OSA

All patients will undergo baseline ophthalmologic examination as part of a regular clinic visit including best-corrected visual acuity, intraocular pressure, slit lamp exam, dilated retinal exam, fluorescein angiography and optical coherence tomography (OCT). Diagnosis of diabetic macular edema will be confirmed with standard domain OCT. Diagnosis of OSA will be confirmed through gold standard of overnight polysomnography.

Data including demographics, ocular history, best corrected visual acuity, IOP, blood sugar control and sleep metrics will be collected. Serum and aqueous fluid samples will be collected at time of first intravitreal injection including VEGF, Placental growth factor, TGFB, ICAM-1,IL-2, IL-3, IL-6, IL-8, IL-10,IL-17, VCAM-1, MCP-1, Epidermal growth factor, Pigment epithelial derived factor (PEDF), Angiotensin 2 and Platelet derived growth factor (PDGF).

Primary outcome:

Levels of cytokine in serum and aqueous humour

Secondary outcome:

Best-corrected visual acuity

Data analysis:

Level of cytokines in serum and aqueous humor in patients with and without OSA will be compared using T test. Statistical significance is defined as p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Type I/II diabetic patients with evidence of diabetic macular edema requiring treatment with anti-VEGF

Exclusion Criteria:

* Contraindications to intravitreal injection including stroke within the past month, ocular or peri-ocular infection, active intraocular inflammation, hypersensitivity to components of the intra-vitreal injection
* Any other retinal or macular pathology such as retinal detachment and age related macular degeneration
* Patients that have taken any systemic immunosuppressive or anti-inflammatory within the past 30 days
* Impaired mental capacity to comply (eg. dementia)
* Pregnant or breastfeeding women

Min Age: 18 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type I/II diabetic patients with diabetic macular edema undergoing first intravitreal injection.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Cytokines | Jan 2018- Mar 2020
  Level of cytokines between patients with and without OSA

CONTACTS AND LOCATIONS:
Locations (1):
- Uptown Eye Speicialists, Brampton, Ontario, Canada